CLINICAL TRIAL: NCT02510664
Title: Promoting Resilience in Youth With Type 1 Diabetes: Pilot of Strengths-Based Family Intervention to Improve Diabetes Outcomes (Diabetes Strengths Study)
Brief Title: Diabetes Strengths Study - Pilot of Provider-delivered Strengths-based Intervention
Acronym: DSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Marisa Hilliard, Assistant Professor of Pediatrics, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-34857; 1K12DK097696 (NIH)
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Type 1 Diabetes
Keywords: Adolescence; Adherence
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): There is no control/comparator group for this pilot study - all participants receive the intervention
  Interventions: Behavioral: Diabetes Strengths Study

INTERVENTIONS:
Behavioral: Diabetes Strengths Study — The intervention consists of: (A) assessing youth and family diabetes strengths and adherence prior to each visit, and (B) training diabetes care providers to tailor their clinical encounters around reinforcing each patient and family's unique "diabetes strengths profile" generated from the strengths and adherence assessments.

SUMMARY:
The purpose of this study is to determine whether a newly developed intervention is feasible and acceptable to adolescents with type 1 diabetes and their families and diabetes care providers, and to evaluate trends in whether the intervention impacts important diabetes outcomes. The intervention involves diabetes care providers discussing and reinforcing individuals' and families' diabetes management strengths during routine, outpatient diabetes care appointments.

DETAILED DESCRIPTION:
The purpose of this study is to pilot test a newly developed strengths-based clinical intervention delivered by diabetes care providers in the context of routine ambulatory diabetes care, designed to promote resilience and support diabetes management among adolescents with type 1 diabetes and their families. The emphasis of the intervention is shifting the tone of clinical encounters for diabetes care to emphasize and reinforce youths' and families' current diabetes strengths and positive diabetes management behaviors. Youth with type 1 diabetes are seen routinely in clinic every 3-4 months, and this intervention will occur at two consecutive clinic visits. The intervention consists of (A) assessing youth and family diabetes strengths and adherence prior to each visit, and (B) training diabetes care providers to tailor their clinical encounters around reinforcing each patient and family's unique "diabetes strengths profile" generated from the strengths and adherence assessments.

Outcome assessments are conducted at baseline (prior to the start of the intervention) and immediately following the conclusion of the intervention (approximately 6-8 months later). The primary outcome is feasibility and acceptability, measured by qualitative feedback from participants and providers, as well as quantification of recruitment and enrollment, provider adherence to intervention protocol, and time to completion. Secondary (exploratory) outcomes include diabetes regimen adherence, glycemic control, family conflict, diabetes burden, diabetes strengths, and satisfaction with the diabetes care provider relationship. Strengths and adherence assessments are also completed prior to the second clinic visit to generate the diabetes strengths profile.

ELIGIBILITY:
Inclusion Criteria:

1. At least one parent of each adolescent, self-identified as the primary caregiver most involved in diabetes care, will also be enrolled with each adolescent participant. When present, secondary caregivers involved in diabetes management will be invited (not required) to participate.
2. Youth type 1 diabetes diagnosis for at least 12 months, to allow ample opportunity for adjustment to diabetes management
3. Youth and parent fluency in written and spoken English because assessment measures are not available in other languages.

Exclusion Criteria:

(1) Presence of a serious mental illness or developmental disability in youth or parent that would impede participation would exclude eligibility.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 172 (Actual)
Dates: Start 2014-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marisa E Hilliard, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants receive informed consent form and a profile of results from two surveys completed during intervention, other participant data not returned to participant
Supporting Information: ICF
Time Frame: Receive informed consent form upon signing, and receive profile of results from 2 intervention surveys at the intervention sessions
Access Criteria: All participants receive informed consent form and survey result profile

REFERENCES:
- [Result] Hilliard ME, Eshtehardi SS, Minard CG, Wheat S, Gunn S, Sanders C, Klenk R, Anderson BJ. Featured Article: Strengths-Based, Clinic-Integrated Nonrandomized Pilot Intervention to Promote Type 1 Diabetes Adherence and Well-Being. J Pediatr Psychol. 2019 Jan 1;44(1):5-15. doi: 10.1093/jpepsy/jsy051. PMID 29982765

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from diabetes clinics at Texas Children's Hospital
Pre-assignment Details: Of 172 individuals (84 parents, 84 adolescents, 4 providers) consented, n=40 (20 parent-adolescent dyads) did not receive the intervention: 18 (9 dyads) transferred care to a provider not trained in intervention, 20 (10 dyads) because their provider retired & insufficient time to reschedule in study period, 2 (1 dyad) due to time constraints
Groups:
- Adolescent: There is no control/comparator group for this pilot study - adolescents and their parent receive the intervention that is delivered by their provider. The Adolescent group completed different sets of questionnaires than the Parent and Provider groups.
  Diabetes Strengths Study: The intervention consists of: (A) assessing youth and family diabetes strengths and adherence prior to each visit, and (B) training diabetes care providers to tailor their clinical encounters around reinforcing each patient and family's unique "diabetes strengths profile" generated from the strengths and adherence assessments.
- Parent: There is no control/comparator group for this pilot study - adolescents and their parent receive the intervention that is delivered by their provider. The Parent group completed different sets of questionnaires than the Adolescent and Provider groups.
  Diabetes Strengths Study: The intervention consists of: (A) assessing youth and family diabetes strengths and adherence prior to each visit, and (B) training diabetes care providers to tailor their clinical encounters around reinforcing each patient and family's unique "diabetes strengths profile" generated from the strengths and adherence assessment.
- Provider: There is no control/comparator group for this pilot study - adolescents and their parent receive the intervention that is delivered by their provider. The Provider group completed different sets of questionnaires than the Adolescent and Parent groups. Diabetes care providers were trained to deliver the intervention and were asked to complete sets of questionnaires at various timepoints.
  Diabetes Strengths Study: The intervention consists of: (A) assessing youth and family diabetes strengths and adherence prior to each visit, and (B) training diabetes care providers to tailor their clinical encounters around reinforcing each patient and family's unique "diabetes strengths profile" generated from the strengths and adherence assessments.
Period: Overall Study
Arm/Group | Adolescent | Parent | Provider
Started (of 84 consented, n=20 did not receive any intervention (see description in Pre-assignment details)) | 84 | 84 | 4
Completed | 64 | 64 | 4
Not Completed | 20 | 20 | 0
Not completed — Transferred Care | 9 | 9 | 0
Not completed — Provider Retired/No Time to Reschedule | 10 | 10 | 0
Not completed — Time Constraints | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Of 84 parents and 84 adolescents consented, n=40 (20 parent-adolescent dyads) did not receive the intervention (reasons stated in Participant Flow section), resulting in data from 64 adolescents and 64 parents at baseline (as well as 4 providers)
Groups:
- Parent: There is no control/comparator group for this pilot study - adolescents and their parent receive the intervention that is delivered by their provider. The Parent group completed different sets of questionnaires than the Adolescent and Provider groups.
  Diabetes Strengths Study: The intervention consists of: (A) assessing youth and family diabetes strengths and adherence prior to each visit, and (B) training diabetes care providers to tailor their clinical encounters around reinforcing each patient and family's unique "diabetes strengths profile" generated from the strengths and adherence assessments
- Total: Total of all reporting groups
Arm/Group | Adolescent | Parent | Provider | Total
Number analyzed (Participants) | 64 | 64 | 4 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: n represents number with complete data to calculate a score. Ages are not reported for Parents and Providers because the data were not collected.
  years
    number analyzed (Participants) | 64 | 0 | 0 | 64
    (all) | 15.0 (1.8) |  |  | 15.0 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: n represents number with complete data to calculate a score. Sex is not reported for Providers because the data were not collected.
  Participants
    number analyzed (Participants) | 64 | 64 | 0 | 128
    Female | 36 | 53 |  | 89
    Male | 28 | 11 |  | 39
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: n represents number with complete data to calculate a score. Race is not reported for Parents and Providers because the data were not collected.
  Participants
    number analyzed (Participants) | 64 | 0 | 0 | 64
    American Indian or Alaska Native | 0 |  |  | 0
    Asian | 4 |  |  | 4
    Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
    Black or African American | 8 |  |  | 8
    White | 44 |  |  | 44
    More than one race | 8 |  |  | 8
    Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants] — Population: n represents number with complete data to calculate a score.
  participants
    United States | 64 | 64 | 4 | 132
Diabetes Strengths and Resilience Measure - Adolescent [Mean (Standard Deviation); unit: units on a scale] — The Diabetes Strengths and Resilience measure is a self-report assessment of positive behaviors related to diabetes resilience for youth with type 1 diabetes, such as perceived competence to manage the demanding diabetes regimen, to adapt to the unpredictability of diabetes, and to seek help and support with diabetes challenges. The scale range from the minimum to maximum possible score is 0-48. A higher value on this scale represents a better outcome. Population: n represents number with complete data to calculate a score.
  units on a scale
    number analyzed (Participants) | 64 | 0 | 0 | 64
    (all) | 37.0 (6.6) |  |  | 37.0 (6.6)
Diabetes Self-Management Profile - Adolescent Self-Report [Mean (Standard Deviation); unit: units on a scale] — Adolescents will complete the youth-report version of the Diabetes Self-Management Profile Self-Report, a self-reported measure of adherence to diabetes regimen, at baseline and follow-up to assess their perceptions of adherence. The version appropriate to the adolescents' current diabetes regimen (conventional insulin regimen, 24 items; or intensive insulin regimen, 24 items) will be administered. The scale ranges from 0-86, with a higher score representing a better outcome. Population: n represents number with complete data to calculate a score.
  units on a scale
    number analyzed (Participants) | 62 | 0 | 0 | 62
    (all) | 52.5 (10.3) |  |  | 52.5 (10.3)
Diabetes Self-Management Profile - Parent-report [Mean (Standard Deviation); unit: units on a scale] — Parents will rate adolescents' adherence to the diabetes regimen using the 24-item Diabetes Self-Management Profile Self-Report. The version appropriate to their child's current diabetes regimen (conventional insulin regimen, 24 items; flexible insulin regimen, 24 items) was administered. The scale ranges from 0-86, with a higher score representing a better outcome. Population: n represents number with complete data to calculate a score.
  units on a scale
    number analyzed (Participants) | 0 | 63 | 0 | 63
    (all) |  | 54.4 (9.2) |  | 54.4 (9.2)
Diabetes Regimen Adherence (Blood Glucose Monitoring Frequency) [Mean (Standard Deviation); unit: checks per day] — Objective measurement of adherence will occur through blood glucose monitoring frequency (a well-accepted surrogate of overall adherence), obtained via blood glucose meter downloads. The average daily frequency will be calculated over the 14 days prior to the assessment at the Baseline visit. Population: n represents number with complete data to calculate a score.
  checks per day
    number analyzed (Participants) | 58 | 0 | 0 | 58
    (all) | 3.6 (1.4) |  |  | 3.6 (1.4)
Glycemic Control (HbA1c) [Mean (Standard Deviation); unit: percentage] — The American Diabetes Association generally recommends an HbA1c target of <7.5% for individuals younger than 18 years. This target varies depending on the individual, but a glycemic goal around this number reduces risk of long-term complications of diabetes. HbA1c values are collected via fingerstick and blood assay at routine diabetes care visits and values will be extracted from the medical record at each clinic visit during the study period. Population: n represents number with complete data to calculate a score.
  percentage
    number analyzed (Participants) | 62 | 0 | 0 | 62
    (all) | 8.56 (1.60) |  |  | 8.6 (1.6)
Problem Areas in Diabetes - Adolescent Self-report [Mean (Standard Deviation); unit: units on a scale] — Problem Areas in Diabetes - Adolescent measures how bothersome day-to-day problems are for adolescents with type 1 diabetes. The scale range of the minimum to maximum possible score is 26-156. A Lower score represent better a outcome. Population: n represents number with complete data to calculate a score.
  units on a scale
    number analyzed (Participants) | 64 | 0 | 0 | 64
    (all) | 68.6 (28.0) |  |  | 68.6 (28.0)
Problem Areas in Diabetes - Parent-report [Mean (Standard Deviation); unit: units on a scale] — Problem Areas in Diabetes - Parent-report measures how bothersome day-to-day problems are for parents of adolescents with type 1 diabetes. The scale range of the minimum to maximum possible score is 26-156. A Lower score represent better a outcome. Population: n represents number with complete data to calculate a score.
  units on a scale
    number analyzed (Participants) | 0 | 64 | 0 | 64
    (all) |  | 71.3 (25.2) |  | 71.3 (25.2)
Diabetes Family Conflict Scale - Revised, Adolescent-report [Mean (Standard Deviation); unit: units on a scale] — The Diabetes Family Conflict Scale - Revised measures the self-reported level of diabetes-specific conflict in families with adolescents with type 1 diabetes. The scale range of the minimum to maximum possible score is 19-57. A lower value represents a better outcome. Population: n represents number with complete data to calculate a score.
  units on a scale
    number analyzed (Participants) | 62 | 0 | 0 | 62
    (all) | 25.5 (5.7) |  |  | 25.5 (5.7)
Diabetes Family Conflict Scale - Revised, Parent-report [Mean (Standard Deviation); unit: units on a scale] — The Diabetes Family Conflict Scale - Revised measures the self-reported level of diabetes-specific conflict in families with adolescents with type 1 diabetes. The scale range of the minimum to maximum possible score is 19-57. A lower value represents a better outcome. Population: n represents number with complete data to calculate a score.
  units on a scale
    number analyzed (Participants) | 0 | 64 | 0 | 64
    (all) |  | 24.7 (4.8) |  | 24.7 (4.8)
Adolescent-provider relationship, adolescent-report [Mean (Standard Deviation); unit: units on a scale] — The adolescent-provider relationship scale measures self-reported feelings about the relationship between the adolescent and their usual diabetes care provider. The scale range of the minimum to maximum possible score is 1-10. A higher score represents a better outcome. Baseline assessment for this measure was collected immediately after the first intervention session. Population: n represents number with complete data to calculate a score
  units on a scale
    number analyzed (Participants) | 62 | 0 | 0 | 62
    (all) | 7.9 (1.6) |  |  | 7.9 (1.6)
Provider-family relationship, provider-report [Mean (Standard Deviation); unit: units on a scale] — The Provider-Family Relationship scale measures the provider's perspective on the quality of their relationship with the teen and family. 4 healthcare providers completed this scale for 60 families. The scale range of the minimum to maximum possible score is 1-10. A higher score represents a better outcome. Baseline assessment for this measure was collected immediately after the first intervention session. Population: n represents number with complete data to calculate a score. 4 healthcare providers completed this scale for 60 families.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 4 | 4
    (all) |  |  | 8.7 (1.0) | 8.7 (1.0)
PedsQL-Healthcare Satisfaction, parent-report [Mean (Standard Deviation); unit: units on a scale] — The PedsQL Healthcare Satisfaction survey measures how happy parents are with their child's healthcare provider in the several categories relevant to the care of type 1 diabetes. An overall mean score is obtained from individual mean scores of 6 sub-scales, which include information, inclusion of family, communication, technical skills, emotional needs, and overall satisfaction. The scale range of the minimum to maximum possible score is 0-100. A higher score represents a better outcome. Population: n represents number with complete data to calculate a score.
  units on a scale
    number analyzed (Participants) | 0 | 63 | 0 | 63
    (all) |  | 96.4 (6.5) |  | 96.4 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Study Design
Description: Measured by percent of recruited families that enrolled in study
Time Frame: Immediately following Enrollment (Baseline)
Population: Over 12 months (10/2014-9/2015), staff screened 212 adolescents for eligibility via electronic medical record, of whom 8 could not be contacted, 11 opted out of learning about research before the study could be introduced, & 88 were ineligible. Of the remaining 105 adolescents, 21 declined to participate, resulting in a consent rate of 80% (n=84).
Measure: Count of Participants; unit: Participants
Groups:
- Parent: There is no control/comparator group for this pilot study - all adolescents and their parents receive the intervention that is delivered by a participating provider. The Parent group completed different sets of questionnaires than the Adolescent and Provider groups.
  Diabetes Strengths Study: The intervention consists of: (A) assessing youth and family diabetes strengths and adherence prior to each visit, and (B) training diabetes care providers to tailor their clinical encounters around reinforcing each patient and family's unique "diabetes strengths profile" generated from the strengths and adherence assessments.
Arm/Group | Adolescent | Parent
Number analyzed (Participants) | 105 | 105
Participants | 84 | 84

2. Primary Outcome: Feasibility of Study Design
Description: Measured by percent of enrolled participants who receive full dose
Time Frame: 6-8 months after enrollment (follow-up timepoint)
Population: 84 ppts enrolled. 64 (76% of consented, 61% of eligible invited to participate) completed baseline surveys & were eligible to participate in the intervention. 63 (75% of consented, 98% of ppts with baseline data) received at least one intervention session. 53 (63% of consented, 83% of ppts with baseline data) completed 2 intervention sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescent | Parent
Number analyzed (Participants) | 84 | 84
Participants | 53 | 53

3. Primary Outcome: Feasibility of Study Design
Description: Measured by time to complete intervention in months since enrollment in study.
Time Frame: 6-8 months after enrollment (follow-up timepoint)
Population: Includes participants who completed post-intervention data
Measure: Mean (Standard Deviation); unit: months since enrollment
Arm/Group | Adolescent | Parent
Number analyzed (Participants) | 63 | 63
months since enrollment | 8.3 (3.6) | 8.3 (3.6)

4. Primary Outcome: Feasibility of Study Design
Description: Measured by percent of participants who provided complete data from all questionnaires.
Time Frame: 6-8 months after intervention begins (immediately following second study visit)
Population: Out of 84 enrolled and 64 who provided baseline data, 60 (71% of enrolled, 94% of ppts with baseline data) provided post-intervention questionnaire battery (some individual measures may not have been complete to calculate a score)
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescent | Parent | Provider
Number analyzed (Participants) | 84 | 84 | 4
Participants | 60 | 60 | 4

5. Primary Outcome: Acceptability: Number of Participants That Felt the Intervention Was Well-Received
Description: The number of participants that felt the intervention was well-received was collected for Adolescents, Parents, and Providers. To determine if the intervention was well-received, verbal responses from qualitative interviews with were coded for types of participant feedback by the study team. We coded these data qualitatively and classified them as Positive, Negative, or Neutral.
Time Frame: 6-8 months after enrollment (follow-up timepoint)
Population: n = number with complete data at this follow-up timepoint to calculate a score.
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescent | Parent | Provider
Number analyzed (Participants) | 53 | 52 | 4
Participants
  Positive | 46 | 44 | 4
  Negative | 0 | 0 | 0
  Neutral | 7 | 8 | 0

6. Secondary Outcome: Diabetes Strengths
Description: Adolescent will self-report on the frequency of 12 resilience-promoting behaviors via the Diabetes Strengths and Resilience, a self-report assessment of positive behaviors related to diabetes resilience for youth with type 1 diabetes, such as perceived competence to manage the demanding diabetes regimen, to adapt to the unpredictability of diabetes, and to seek help and support with diabetes challenges. The scale ranges from 0-48, with a higher score representing a better outcome.
Time Frame: 3-4 months after enrollment (mid-intervention timepoint), and 6-8 months after enrollment (follow-up timepoint)
Population: n = number with complete data at baseline to calculate a score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adolescent
Number analyzed (Participants) | 64
units on a scale
  3-4 months after enrollment (mid-intervention): number analyzed (Participants) | 53
  3-4 months after enrollment (mid-intervention) | 38.1 (5.6)
  6-8 months after enrollment (follow-up timepoint): number analyzed (Participants) | 61
  6-8 months after enrollment (follow-up timepoint) | 39.7 (5.8)

7. Secondary Outcome: Diabetes Self-Management Profile - Parent-report
Description: Parents will rate adolescents' adherence to the diabetes regimen using the 24-item Diabetes Self-Management Profile Self-Report. The version appropriate to their child's current diabetes regimen (conventional insulin regimen, 24 items; flexible insulin regimen, 24 items) was administered. The scale ranges from 0-86, with a higher score representing a better outcome.
Time Frame: 3-4 months after enrollment (mid-intervention timepoint), and 6-8 months after enrollment (follow-up timepoint)
Population: n = number with complete data at baseline timepoint to calculate a score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent
Number analyzed (Participants) | 63
units on a scale
  3-4 months after enrollment (mid-intervention): number analyzed (Participants) | 53
  3-4 months after enrollment (mid-intervention) | 55.2 (9.5)
  6-8 months after enrollment (follow-up timepoint): number analyzed (Participants) | 59
  6-8 months after enrollment (follow-up timepoint) | 56.9 (10.0)

8. Secondary Outcome: Diabetes Self-Management Profile - Adolescent-report
Description: Adolescents will complete the youth-report version of the Diabetes Self-Management Profile Self-Report, a self-reported measure of adherence to diabetes regimen, at baseline and follow-up to assess their perceptions of adherence. The version appropriate to the adolescents' current diabetes regimen (conventional insulin regimen, 24 items; or intensive insulin regimen, 24 items) will be administered. The scale ranges from 0-86, with a higher score representing a better outcome.
Time Frame: 6-8 months after enrollment (follow-up timepoint)
Population: n = number with complete data at this follow-up timepoint to calculate a score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adolescent
Number analyzed (Participants) | 59
units on a scale | 56.9 (10.1)

9. Secondary Outcome: Diabetes Regimen Adherence (Blood Glucose Monitoring Frequency)
Description: Objective measurement of adherence will occur through blood glucose monitoring frequency (a well-accepted surrogate of overall adherence), obtained via blood glucose meter downloads. The average daily frequency will be calculated over the 14 days prior to the assessment at the Baseline and second study visits.
Time Frame: 6-8 months after enrollment (follow-up timepoint)
Population: n = number with complete meter data at this follow-up timepoint to calculate a score
Measure: Mean (Standard Deviation); unit: checks per day
Arm/Group | Adolescent
Number analyzed (Participants) | 53
checks per day | 3.64 (1.36)

10. Secondary Outcome: Glycemic Control
Description: Diabetes is typically diagnosed with an HbA1c of 6.5% or higher. At the time of this study, the American Diabetes Association generally recommended an HbA1c target of <7.5% for individuals younger than 18 years (the specific target varies depending on the individual). The DCA 2000 HbA1c Analyzer (Siemens-Bayer) was used for point of care HbA1c analysis, it has an analytical measurement range for HbA1c of 2.5% to 14.0%. HbA1c values are collected via fingerstick and blood assay at routine diabetes care visits and values will be extracted from the medical record at each clinic visit during the study period.
Time Frame: 6-8 months after enrollment (follow-up timepoint)
Population: n = number with HbA1c value available at this follow-up timepoint
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Adolescent
Number analyzed (Participants) | 59
percentage | 8.54 (1.59)

11. Secondary Outcome: Problem Areas in Diabetes - Teen
Description: Burden will be assessed via the Problem Areas in Diabetes - Teen. The scale has 26 items and demonstrates good psychometric properties. The scale ranges from 26-156, with higher scores representing worse outcomes.
Time Frame: 6-8 months after enrollment (follow-up timepoint)
Population: n = number with complete data at this follow-up timepoint to calculate a score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adolescent
Number analyzed (Participants) | 61
units on a scale | 61.6 (23.6)

12. Secondary Outcome: Diabetes Burden - Problem Areas in Diabetes - Parent-report
Description: Burden will be assessed via the Problem Areas in Diabetes measures for parents. The scale has 26 items and demonstrates good psychometric properties. The scale ranges from 26-156, with a higher score representing a worse outcome.
Time Frame: 6-8 months after enrollment (follow-up timepoint)
Population: n = number with complete data at this timepoint to calculate a score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent
Number analyzed (Participants) | 59
units on a scale | 64.6 (20.3)

13. Secondary Outcome: Diabetes-related Family Conflict (Parent-report)
Description: Parents will complete the Diabetes Family Conflict Scale Revised, a 19 item scale with good reliability and validity. The scale ranges from 19-57, with higher scores representing a worse outcome.
Time Frame: 6-8 months after enrollment (follow-up timepoint)
Population: n = number with complete data at this follow-up timepoint to calculate a score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent
Number analyzed (Participants) | 58
units on a scale | 24.9 (4.6)

14. Secondary Outcome: Diabetes-related Family Conflict (Adolescent Report)
Description: Adolescents will also complete the Diabetes Family Conflict Scale Revised, a 19 item scale with good reliability and validity. The scale ranges from 19-57, with higher scores representing a worse outcome.
Time Frame: 6-8 months after enrollment (follow-up timepoint)
Population: n = number with complete data at this follow-up timepoint to calculate a score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adolescent
Number analyzed (Participants) | 60
units on a scale | 24.3 (4.8)

15. Secondary Outcome: Healthcare Satisfaction - PedsQL Healthcare Satisfaction Parent-report
Description: To assess healthcare satisfaction, parents will complete three subscales of the PedsQL Inventory Healthcare Satisfaction Generic Module, assessing their satisfaction with communication, inclusion of family, and how well the patient's emotional needs are addressed during the clinical encounter (13 items). The scale ranges from 0-100, with a higher score representing a better outcome.
Time Frame: 6-8 months after enrollment (follow-up timepoint)
Population: n = number with complete data at this follow-up timepoint to calculate a score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent
Number analyzed (Participants) | 59
units on a scale | 96.1 (10.3)

16. Secondary Outcome: Adolescent-provider Relationship - Adolescent-report
Description: Adolescents will rate their overall satisfaction with the patient-provider relationship on a 1-10 scale single item developed for this study, as there is no validated youth-report measure of satisfaction with care. The scale ranges from 1-10, with higher scores representing a better outcome.
Time Frame: 6-8 months after enrollment (follow-up timepoint)
Population: n = number with data at this follow-up timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adolescent
Number analyzed (Participants) | 56
units on a scale | 8.5 (1.8)

17. Secondary Outcome: Provider-family Relationship, Provider-report
Description: Providers will rate their overall satisfaction with the provider-family relationship on a scale developed for this study. The Provider-Family Relationship scale measures the provider's perspective on the quality of their relationship with the teen and family. 4 healthcare providers completed this scale for 48 families. The scale range of the minimum to maximum possible score is 1-10. A higher score represents a better outcome.
Time Frame: 6-8 months after enrollment (follow-up timepoint)
Population: n represents number with complete data to calculate a score. 4 healthcare providers completed this scale for 48 families (adolescent-parent dyads).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Provider
Number analyzed (Participants) | 48
units on a scale | 9.1 (1.0)

ADVERSE EVENTS:
Arm/Group | Adolescent | Parent | Provider
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/84 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/84 | 0/4
Other Adverse Events (participants affected / at risk) | 0/84 | 0/84 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT02510664/Prot_SAP_000.pdf